CLINICAL TRIAL: NCT03403673
Title: Clinical Frailty Scale Validation in Patients Scheduled for Vascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South Tees Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2016053
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Frailty assessment tools — There is evidence to suggest that patients who are frail have a higher risk of developing complications after major surgery. Our aim is to ask you simple questions about your physical ability to perform daily life activities, assess your general health condition and ask you to do simple tasks such as drawing a clock or walking for a short distance to assess your speed of walking. Our main aim is to identify a tool that will assist us to identify patients who are at risk of frailty

SUMMARY:
Major vascular operations put the body under stress. We are trying to find out if the general health of a patient and the stress resulting from surgery can lead to the development of complications after surgery as well as increase the length of time spent in hospital.

There is evidence to suggest that patients who are frail have a higher risk of developing complications after major surgery.

Our aim is to ask you simple questions about your physical ability to perform daily life activities, assess your general health condition and ask you to do simple tasks such as drawing a clock or walking for a short distance to assess your speed of walking. Our main aim is to identify a tool that will assist us to identify patients who are at risk of frailty.

ELIGIBILITY:
Inclusion Criteria: Patients attending vascular pre assessment clinic Age > 60 -

Exclusion Criteria: Refusal or inability to provide informed consent. Patients under 60 years of age. Patients not undergoing a vascular procedure.

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All vascular patients attending the preoperative assessment clinics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Clinical frailty scale validation in preoperative assessment of patients scheduled for vascular surgery | June 2018
  Identify a tool that will assist us to identify patients who are at risk of frailty.

CONTACTS AND LOCATIONS:
Locations (1):
- South Tees Hospitals NHS Foundation Trust, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ayyash R, Knight J, Kothmann E, Eid M, Ayyash K, Colling K, Yates D, Mill A, Danjoux G. Utility and reliability of the Clinical Frailty Scale in patients scheduled for major vascular surgery: a prospective, observational, multicentre observer-blinded study. Perioper Med (Lond). 2022 Jan 31;11(1):6. doi: 10.1186/s13741-022-00240-9. PMID 35101117